CLINICAL TRIAL: NCT02134535
Title: Optimization of the ex Vivo Challenge
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Katherine Bunge, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO13120447
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Optimization of Laboratory Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- laboratory specimens: cervical biopsies vaginal biopsies blood

SUMMARY:
The overall purpose of this research study is to collect vaginal and cervical biopsies from healthy HIV negative participants. These samples will enable investigators to optimize laboratory methods and explore implementation challenges associated with the ex vivo challenge model. The first objective is to assess which HIV virus is best for use in the model. The second objective is to determine the best endpoint for the assay.

The primary aim of this study is to collect an adequate number of cervical and vaginal biopsies to support the optimization of an ex vivo challenge model. This ex vivo challenge model has been and will continue to be used in topical microbicide clinical trials to predict the efficacy of candidate drugs.

DETAILED DESCRIPTION:
The development of surrogates to predict HIV prevention product safety and efficacy is a high priority. An ex vivo challenge model is one such promising surrogate. Colonic tissue exposed to rectally applied microbicides in vivo and then challenged with HIV in the lab showed significant reduction in HIV replication when compared to tissue exposed to placebo gel. Currently, the ex vivo challenge model for ectocervical and vaginal tissue is being developed at the Dezzutti lab at the Magee Womens Research Institute in Pittsburgh, PA. Questions which need to be addressed in order to optimize the model include which HIV virus is most appropriate to use to challenge the tissue, is qPCR a more appropriate endpoint and marker of infection, and can frozen tissue perform as well as fresh tissue in the challenge model.

In this study, we will collect vaginal and cervical biopsies to use in the optimization of laboratory procedures. We will obtain the sample(s) from healthy HIV negative women. Samples will be collected and taken to Magee-Womens Research Institute as laboratory specimens. Written consent will be obtained by an investigator or co-investigator prior to the collection of any samples.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45
2. Free from abnormal vaginal discharge or other current vaginal symptoms
3. HIV uninfected. Note: if a woman recently participated in a recent research study and has an HIV test result available from that study, this will suffice provided the date of the test is within 6 months of the enrollment visit for this trial. Otherwise, the potential participant should under go testing at the first study visit.
4. Willing and able to give informed consent to take place in the study
5. Willing to undergo a pelvic examination and genital biopsies
6. Willing to provide contact information
7. Agree to be sexually abstinent for two weeks beginning one week prior to the enrollment visit

Exclusion Criteria:

1. Menopausal
2. Pregnant or within 90 days of last pregnancy
3. Hysterectomy
4. Use of a diaphragm, NuvaRing or spermicide for contraception
5. Reports a course of antibiotic therapy in the 14 days prior to enrollment
6. Known history of platelet disorder or coagulapathy.
7. Participation in another microbicide or contraceptive study or a study involving cervical and/or vaginal biopsies within one month of enrollment
8. Use of any spermicide or spermicide-lubricated condom within one week of enrollment.
9. Use of any internal vaginal device or product with the exception of tampons within one week of enrollment
10. Any other condition that in the opinion of the site investigator would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, non-pregnant, HIV negative women
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
cervical biopsy | Day 1
vaginal biopsy | Day 1

SECONDARY OUTCOMES:
blood draw | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Bunge, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States